CLINICAL TRIAL: NCT04603950
Title: IPICK Blocking for Extension Recovery in TKA With Preoperative Moderate Flexion Contracture
Brief Title: IPICK Blocking for TKA With Moderate Flexion Contracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QiXin2
Record Dates: First submitted 2020-10-08; First posted 2020-10-27 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis; Flexion Contracture of Knees; Anesthesia, Local
Keywords: IPACK; knee osteoarthritis; Flexion Contracture of Knees
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): The first 20 patients received Continue Adductor Canal Block + Infiltration between the Popliteal Artery and Capsule of the Knee
  Interventions: Procedure: CACB+IPACK
- control group (Sham Comparator): The second 20 patients received Continue Adductor Canal Block alone
  Interventions: Procedure: CACB

INTERVENTIONS:
Procedure: CACB+IPACK — continue adductor canal block plus Infiltration between the Popliteal Artery and Capsule of the Knee
  Arms: study group
Procedure: CACB — continue adductor canal block
  Arms: control group

SUMMARY:
Clinical effect of intermittent multiple IPICK blocking on TKA for knee osteoarthritis with flexion contracture between 5 ° and 10 °

DETAILED DESCRIPTION:
From October 2020 to January 2021, 40 knee osteoarthritis patients with flexion contracture between 5 ° and 10 ° total knee arthroplasty are enrolled in this study. 20 patients are treated with Adductor Canal Block + Infiltration between the Popliteal Artery and Capsule of the Knee, and 20 patients are treated with Adductor Canal Block alone.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis was knee osteoarthritis
2. The flexion contracture was between 5 and 10 degrees
3. ASA grade I-III

Exclusion Criteria:

1. Lower extremity neuropathy.
2. Contraindications of nerve anesthesia or regional anesthesia.
3. unable to cooperate, allergic to the drugs used in this study.
4. Non steroidal anti-inflammatory drugs are not tolerated.
5. chronic opioid consumption (daily or almost daily use)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
evaluation of pain | 6 hours after surgery
  Visual Analog Score for pain at rest, straightening, flexion at 45 ° and walking, the minimum and maximum values are 0 to 10, higher scores mean a worse outcome.
evaluation of pain | postoperative day 1
  Visual Analog Score for pain at rest, straightening, flexion at 45 ° and walking, the minimum and maximum values are 0 to 10, higher scores mean a worse outcome.
evaluation of pain | postoperative day 2
  Visual Analog Score for pain at rest, straightening, flexion at 45 ° and walking, the minimum and maximum values are 0 to 10, higher scores mean a worse outcome.
evaluation of pain | postoperative day 3
  Visual Analog Score for pain at rest, straightening, flexion at 45 ° and walking, the minimum and maximum values are 0 to 10, higher scores mean a worse outcome.
extension angle | before surgery
  degree of the extension of knee
extension angle | 0 hour after surgery
  degree of the extension of knee
extension angle | 6 hour after surgery
  degree of the extension of knee
extension angle | postoperative day 1
  degree of the extension of knee
extension angle | postoperative day 2
  degree of the extension of knee
extension angle | postoperative day 3
  degree of the extension of knee

SECONDARY OUTCOMES:
range of motion | 6 hour after surgery
  degree of range of motion from extension to flexion of knee
range of motion | postoperative day 1
  degree of range of motion from extension to flexion of knee
range of motion | postoperative day 2
  degree of range of motion from extension to flexion of knee
range of motion | postoperative day 3
  degree of range of motion from extension to flexion of knee
opioid consumption | through hospitalization, an average of 7 days
  total opioid consumption measured by milliliter.
nerve block related symptoms | through hospitalization, an average of 7 days
  the incidence of numbness of the nerve related skin
postoperative acute pain | through hospitalization, an average of 7 days
  number of cases whose Visual Analog Score for pain was more than 5

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: No